CLINICAL TRIAL: NCT04147078
Title: Adjuvant Treatment in Cancer Patients with Neoantigen-primed DC Vaccine : a Single-arm, Open-label, Prospective Clinical Trial
Brief Title: Personalized DC Vaccine for Postoperative Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Department of Medical Oncology, Cancer Center, West China Hospital, Sichuan University, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHANT-191
Record Dates: First submitted 2019-08-24; First posted 2019-10-31 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer; Hepatocellular Carcinoma; Non-Small-Cell Lung Cancer; Colon Rectal Cancer
Keywords: Cell therapy; safety; clinical efficacy; adjuvant treatment; locally advanced cancer
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cell_therapy (Experimental): tumor neoantigen primed DC vaccines are administrated, 2-3 week interval, totally 3-5 times
  Interventions: Biological: DC vaccine subcutaneous administration

INTERVENTIONS:
Biological: DC vaccine subcutaneous administration — subcutaneous administration

SUMMARY:
The study is aimed to the test efficacy and safety of neoantigen-primed dendritic cell (DC) cell vaccine therapy for postoperative locally advanced gastric cancer, hepatocellular carcinoma, lung cancer and colorectal cancer, and to explore the biomarkers related to efficacy and adverse event.

DETAILED DESCRIPTION:
Postoperative patients with pathological confirmed locally advanced gastric cancer, hepatocellular carcinoma, non-small cell lung cancer and colorectal cancer with standard adjuvant treatment are enrolled. This is a prospective exploratory trial. Patients' tumor tissues are subsequent to whole exosome sequencing and possible neoantigens are identified. DC is in vitro primed with synthesized peptides. Both adverse events and responses are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a first diagnosis of gastric cancer, hepatocellular carcinoma, non-small cell lung cancer, colorectal cancer who have undergone a curative resection or ablation
* Anticipated life time > 3month
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Adequate organ functions

Exclusion Criteria:

* Any evidence of tumor metastasis or co-existing malignant disease
* Tumor emergency
* Abnormal coagulation condition
* Contagious diseases, such as hepatitis B virus, hepatitis C virus, human immunodefficiency virus, tuberculosis infection
* Concomitant tumors
* Immunological co-morbidities

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | Up to 5 years
  Defined as the time from the surgery to the first documented disease recurrence or death (by any cause), whichever occurs first

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 10 years
  Defined by the time between the date of randomization and the date of death
Incidence of Treatment-Related Adverse Events [Safety and Tolerability] | 3 months after the last administration of cells
  Defined by treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Qiu Li, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No